CLINICAL TRIAL: NCT01390714
Title: An Open-label, Cross-over, Pharmacodynamic and Pharmacokinetic Study of E3710 Following Oral Administration to Healthy, Male, Japanese Subjects
Brief Title: Pharmacodynamic and Pharmacokinetic Study of E3710 Following Oral Administration to Healthy, Male, Japanese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: E3710-A001-003
Record Dates: First submitted 2011-06-28; First posted 2011-07-11 (Estimated); Last update posted 2012-03-14 (Estimated); Status verified 2012-03

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: Proton Pump Inhibitors; Gastroesophageal Reflux Disease; pharmacokinetics; pharmacodynamics
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — 2-(4-(2,2-dimethyl-1,3-dioxan-5-yl)methoxy-3,5-dimethylpyridin-2-yl)methylsulfinyl-1H-benzimidazole

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: E3710
- 2 (Experimental)
  Interventions: Drug: E3710

INTERVENTIONS:
Drug: E3710 — Arm A:
  1. E3710 40 mg→RPZ 10 mg→E3710 20 mg
  2. RPZ 10 mg→E3710 20 mg→E3710 40 mg
  3. E3710 20 mg→E3710 40 mg→RPZ 10 mg
  Crossover study of E3710 40 mg, E3710 20 mg, and PRZ 10 mg, once daily, for 5 days, oral administration.
  Arms: 1
Drug: E3710 — Arm B:
  1. E3710 40 mg→E3710 80 mg→EPZ 40 mg
  2. E3710 80 mg→EPZ 40 mg →E3710 40 mg
  3. EPZ 40 mg→E3710 40 mg→E3710 80 mg
  Crossover study of E3710 40 mg, E3710 80 mg, and EPZ 40 mg, once daily, for 5 days, oral administration.
  Arms: 2

SUMMARY:
The purpose of this study is to investigate the pharmacodynamics (PD) and pharmacokinetics of E3710 following oral administration to Healthy Male Japanese Subjects

DETAILED DESCRIPTION:
This study will be conducted in healthy, male, Japanese subjects using an open-label, randomized, crossover design with comparison under multiple oral doses of E3710. Rabeprazole or Esomeprazole will be used in this study as marketed comparators. In each arm, pharmacodynamics will be measured in regard to intragastric pH. The measurements will be recorded using a pH probe with esophageal measurement capability for 24 hours post-dose. Pharmacokinetics measurements will also be conducted in all dosing stages for collecting serial blood samples.

ELIGIBILITY:
Inclusion Criteria

1. Subjects who received a full explanation about objectives and contents of this study and provided written consent to participate in this study by their own free will before the start of screening.
2. Japanese, healthy, male adults, 20-40 years of age on the day of consent.
3. Japanese subjects must be first generation Japanese (born in Japan of Japanese parents and Japanese grandparents), must have lived no more than 5 years outside of Japan and must not have changed their life style or habits, including diet, while living outside of Japan.
4. CYP2C19 homo or heterozygous extensive metabolizers.
5. Subjects who have no current infection with Helicobacter pylori (H. pylori).
6. Subjects with body mass index (BMI) 18.5-25.0 kg/m2 at the time of screening.
7. Subjects who received screening examination within 4 weeks before entering the Phase I unit in Stage 1 and were judged to be eligible for this study by the investigator.

Exclusion Criteria

1. Likely allergy or sensitivity to any components of E3710 based on known allergies to drugs of the same class (e.g. proton pumps inhibitors, specifically RPZ or EPZ) or which in the opinion of the Principal Investigator might increase the potential for adverse events.
2. Subjects with present or previous history of drug allergy, food allergy or clinically problematic allergy (e.g. chronic asthma or urticaria).
3. Subjects with diseases that may affect evaluation of the study drug such as gastrointestinal, hepatic, renal, respiratory, endocrine, blood, nervous, mental or cardiac vascular diseases or congenital metabolic disorders at the time of screening or within 4 weeks before hospitalization in each stage of the study.
4. Subjects with history of surgical therapies (such as resection of the liver, the kidney or the digestive tracts) that may influence pharmacokinetics of the study drug.
5. Subjects who had 10% or more of body weight changes during a period from screening to Day 1 of hospitalization in each stage of the study.
6. Subjects who had beverages containing caffeine (such as coffee, tea, chocolate or cola) within 72 hours before hospitalization in each stage of the study.
7. Subjects who had grapefruit juice or food and drinks containing grapefruit within 72 hours before hospitalization in each stage of the study.
8. Subjects who had alcoholic beverages within 72 hours before hospitalization in each stage of the study.
9. Subjects who cannot quit smoking during hospitalization.
10. Subjects who performed vigorous exercise or hard labor (more than 1 hour in a day or 5 days or more in a week) within 2 weeks before hospitalization in each stage of the study.
11. Subjects who are found to have abnormal clinical symptoms or organ function disorders requiring medical treatment in examinations of medical history, symptoms and signs, vital signs, ECG or laboratory tests.
12. Subjects with QTC longer than 450 msec in 12-lead electrocardiography (Bazett's method).
13. Subjects with history of alcohol or drug abuse, who are suspected to have such the history or who have positive reaction in urinary drug test at the time of screening or hospitalization of the study.
14. Subjects who used any ethical drugs within 4 weeks before hospitalization in each stage of the study *.
15. Subjects who took any OTC drugs (including PPIs and H2-receptor antagonists), antacids, nutrients, vitamin preparations or preparations containing herb (including Chinese medicines and food products) within one week before hospitalization in each stage of the study. However, for the herb preparations, which are known to induce cytochrome P450, drug metabolizing enzyme (e.g. preparations and food products containing St. John's wort), subjects who took such the preparations within 4 weeks before hospitalization in each stage of the study.
16. Subjects who used any other investigational drugs or investigational medical equipment within 16 weeks before hospitalization in each stage of the study.
17. Subjects who received blood transfusions within 12 weeks before hospitalization in each stage of the study, or who donated 400 mL or more of whole blood within 12 weeks or 200 mL or more of whole blood within 4 weeks before hospitalization in each stage of the study.
18. Subjects who had any infections requiring medical treatments within 4 weeks before hospitalization in each stage of the study.
19. Subjects who are positive for hepatitis B surface antigen (HBs antigen), hepatitis C virus (HCV) antibody or qualitative test for syphilis.
20. Subjects who were diagnosed as acquired immunodeficiency syndrome (AIDS) or who had positive reaction for human immunodeficiency virus (HIV).
21. Subjects who are not willing to observe the rules of this study or who cannot observe them.
22. Patients who were judged to be inappropriate for participation in this study by the investigator or subinvestigator. *: Excluding drugs prescribed by the investigator in case of necessity for treatment of adverse events after hospitalization.

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2011-07; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Pharmacodynamic effect by ph monitoring will be evaluated. | Day 1 and Day 5
  Summary statistics of the measurements and changes from pre-dose values to post-dose values of intragastric pH 1-, pH 2-, pH 3-, pH 4-, pH 5-, and pH 6 holding time, mean of the intragastric pH and median of intragastric pH are to be calculated by dose. In addition, the mean and median intragastric pH for the hours 1-14 and 14-24 (8:00-22:00 and 22:00-8:00) should be calculated for baseline and each pH-recording period.
Pharmacokinetics parameters Cmax will be calculated. | 4 weeks
  Summary statistics of E3710/RPZ/EPZ pharmacokinetic parameters on Day 1 and Day 5 of administration are to be calculated by dose. Relationship of Cmax to dose of E3710 is to be examined.
Pharmacokinetics parameter AUC will be calculated. | 4 weeks
  Summary statistics of E3710/RPZ/EPZ pharmacokinetic parameters on Day 1 and Day 5 of administration are to be calculated by dose. Relationship of AUC to dose of E3710 is to be examined.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Yen, Principal Investigator — California Clinical Trials
Locations (1):
- Glendale, California, United States